CLINICAL TRIAL: NCT04095793
Title: A Phase 3, 182-week, Open-Label, Extension Study to Investigate the Safety and Tolerability of TD-9855 in Treating Symptomatic Neurogenic Orthostatic Hypotension (Symptomatic nOH) in Subjects With Primary Autonomic Failure
Brief Title: Phase 3 Open-Label Extension Study of TD-9855 for Treating Symptomatic nOH in Subjects With Primary Autonomic Failure
Acronym: OAK
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Stopped early due to company decision. Company decision based on analysis results in TD-9855-0169.
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0171; 2019-002425-30 (EudraCT Number)
Record Dates: First submitted 2019-08-01; First posted 2019-09-19 (Actual); Results first posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Symptomatic Neurogenic Orthostatic Hypotension
Keywords: Symptomatic Neurogenic Orthostatic Hypotension; sympomatic nOH; multiple symptom atrophy; MSA; Parkinson's disease; PD; pure autonomic failure; PAF; orthostatic hypotension; OH; ampreloxetine; 171; low blood pressure; dizziness; fainting; blacking out; lightheadedness; norepinephrine; hypotension; OAK
MeSH Terms: conditions — Parkinson Disease; Pure Autonomic Failure; Hypotension, Orthostatic; Hypotension; Dizziness; Syncope | interventions — ampreloxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ampreloxetine (Experimental): Participants will receive a single, oral, daily dose of active drug (TD-9855) for 182 weeks.
  Interventions: Drug: ampreloxetine

INTERVENTIONS:
Drug: ampreloxetine — Oral tablet, QD
  Other Names: TD-9855

SUMMARY:
A Phase 3, multi-center, open-label study to evaluate the safety and tolerability of ampreloxetine in subjects with primary autonomic failures (MSA, PD, and PAF) and symptomatic nOH over 182 weeks.

DETAILED DESCRIPTION:
This is a Phase 3, multi-center, open-label study to evaluate the safety and tolerability of ampreloxetine in subjects with primary autonomic failures (MSA, PD, and PAF) and symptomatic nOH. The study consists of 3 periods: (i) 26-week treatment, (ii) 156-week treatment extension, and (iii) 2-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Completion of Study 0170 and, in the opinion of the Investigator, would benefit from long-term treatment with ampreloxetine.
* The subject must be able to understand the nature of the study and must provide written informed consent prior to the conduct of any study procedures (including any changes occurring in the subject's current therapeutic regimen).
* The subject must be willing to continue on treatment and must continue to meet all the inclusion criteria for the preceding study (Study 0170) except, a score of >4 in OHSA#1.

Exclusion Criteria:

* Subjects may not be enrolled in another clinical trial.
* Psychiatric, neurological, or behavioral disorders that may interfere with the ability of subjects to give informed consent, or interfere with the conduct of the study.
* Medical, laboratory, or surgical issues deemed by the Investigator to be clinically significant.
* Hypersensitivity to ampreloxetine or the formulation excipients.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2021-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (55):
- United States (13):
  - Colorado Springs Neurological Associates, Colorado Springs, Colorado
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Neurostudies, Inc., Port Charlotte, Florida
  - Rush University Medical Center, Chicago, Illinois
  - NorthShore University HealthSystem, Glenview, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - New York University School of Medicine, New York, New York
  - University of Cincinnati Medical Center (UCGNI), Cincinnati, Ohio
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Inland Northwest Research, Spokane, Washington
- Australia (3):
  - Concord Hospital, Neurosciences Department, Concord, New South Wales
  - Clinical Trials Centre, Level 3 Monash Health Translational Precinct Building Monash Medical Centre, Clayton, Victoria
  - Perron Institute for Neurological and Translational Science, Nedlands, Western Australia
- Universitätsklinikum Tulln Abteilung fur Neurologie, Tulln, Austria
- Bulgaria (2):
  - MHATNP -Sv. Naum- EAD, Sofia
  - MHATNP Sv. Naum EAD Clinic of Neurological Diseases for Locomotor Disorders, Sofia
- Montreal Neurological Institute & Hospital, Montreal, Quebec, Canada
- Bispebjerg Hospital, Copenhagen, Denmark
- Tartu University Hospital, Tartu, Estonia
- CHU de Nîmes - Hôpital Caremeau, Nîmes, Gard, France
- Germany (2):
  - Praxis Dr. med. Christian Oehlwein, Gera, Thuringia
  - Charite - Campus Virchow- Klinikum, Klinik fur Neurologie, Berlin
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Italy (7):
  - Ospedaliera Santa Maria Terni, Terni, Umbria
  - Universita di Bologna-Clinica Neurologica-Dipartimento di Scienze Neurologiche Ospedale Bellaria, Bologna
  - UO Farmacia Centralizzata OM (SC) Ospedale Maggiore, Bologna
  - Fondazione IRCCS CA Granda Ospedale Maggiore Pliclinico - U.O. Neurologia, Milan
  - Fondazione PTV - Policlinico Tor Vergata I U.0.C. Neurologia, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS / Istituto di Neurologia - Ambulatorio Disturbi del Movimento, Roma
  - AOU San Giovanni di Dio e Ruggi d'Aragona, Salerno
- New Zealand Brain Research Institute, Christchurch, New Zealand
- Poland (6):
  - Specjalistyczna Praktyka Lekarska prof.Grzegorz Opala, Katowice
  - Krakowska Akademia Neurologii Sp z o.o. Centrum Neurologii Klinicznej, Krakow
  - Instytut Zdrowia Dr Boczarska-Jedynak SP. Z 0.0., SP. K., Oświęcim
  - Neuro-Care Sp. z o.o. sp. Komandytowa, Siemianowice Śląskie
  - ETG Warszawa, Warsaw
  - Specjalistyczn.e Gabinety Sp. Z o.o., Warsaw
- Campus Neurologico Senior, Torres Vedras, Portugal
- Russia (6):
  - Federal State Budgetary Institution Federal Sibirian Scientific and Clinical Center of Federal Medico-Biological Agency, Krasnoyarsk
  - Federal Sibirian Scientific and Clinical Center of Federal Medico-Biological Agency, Krasnoyarsk
  - SBEI APE Russian Medical Academy of Postgraduate Education of the MoH of the RF, Moscow
  - Limited Liability Company City Neurological Center Sibneiromed, Novosibirsk
  - State Budgetary Institution of Healthcare of Novosibirsk region City Clinical Hospital No. 34, Novosibirsk
  - FSBI "National Medical Research Centre of psychiatry and neurology named after V.M. Bekhterev" of the MOH of the Russian Federation, Saint Petersburg
- Spain (3):
  - Hospital del Mar, Barcelona
  - Hospital de Cruces, Bilbao
  - Hospital Universitario de La Princesa, Madrid
- Ukraine (3):
  - Municipal Instituion of Health: Kharkiv Public Outpatient Clinic 9, Kharkiv Medical Academy of Post-Graduate Education, Department of General Practice - Family Medicine, Kharkiv
  - Lviv Regional Clinical Hospital, Lviv
  - CNE Acad O.I. Yushchenko Vinnytsia Reg Psychoneurological Hospital of Vinnytsia Regional Council, Department of Neurology, Vinnytsia
- United Kingdom (2):
  - The National Hospital for Neurology & Neurosurgery, London, Greater London
  - Re:Cognition Health Ltd, London

IPD SHARING:
Plan to Share IPD: No
Theravance Biopharma, Inc. will not be sharing individual de-identified participant data or other relevant study documents.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 110 participants who completed Study 0170 rolled over into Study 0171. The study was performed in Europe, Asia/Pacific, and the United States between 19 September 2019 and 12 November 2021.
Pre-assignment Details: The study was planned to consist of 3 periods: 26-week treatment,156-week treatment extension, and 2-week follow-up.
Groups:
- Ampreloxetine: Participants received a single dose of 10 mg ampreloxetine once daily (QD) for a planned duration of up to 182 weeks.
Period: Overall Study
Arm/Group | Ampreloxetine
Started | 110
Completed | 0
Not Completed | 110
Not completed — Adverse Event | 3
Not completed — Study Terminated by Sponsor | 103
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Population: The safety analysis set was defined as all enrolled participants who have received at least one dose of ampreloxetine in this study.
Groups:
- Ampreloxetine: Participants received a single dose of 10 mg ampreloxetine QD for a planned duration of up to 182 weeks.
Arm/Group | Ampreloxetine
Number analyzed (Participants) | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (8.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 105
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 108
  More than one race | 0
  Unknown or Not Reported | 0
Primary Diagnosis [Count of Participants; unit: Participants]
  Multiple System Atrophy | 34
  Parkinson's Disease | 58
  Pure Autonomic Failure | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a patient or clinical study participant administered a pharmaceutical product that does not necessarily have to have a causal relationship with this treatment. A TEAE was defined as any AE that begins on or after the date of first dose of study drug up to the date of last dose of study drug plus the number of days in the follow-up period.
  Clinically significant abnormalities in physical and neurological examinations, vital signs, resting 12-lead electrocardiograms, and clinical laboratory evaluations, in addition to incidence of fall, suicidal ideation, and suicidal behavior, were reported as AEs.
Time Frame: Day 1 up to a maximum of 749 days
Population: The safety set was defined as all enrolled participants who received at least 1 dose of ampreloxetine in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Ampreloxetine
Number analyzed (Participants) | 110
Participants | 61

ADVERSE EVENTS:
Time Frame: Day 1 up to a maximum of 749 days
Description: The safety set was defined as all enrolled participants who received at least 1 dose of ampreloxetine in the study.
Arm/Group | Ampreloxetine
All-Cause Mortality (participants affected / at risk) | 1/110
Serious Adverse Events (participants affected / at risk) | 14/110
Other Adverse Events (participants affected / at risk) | 24/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ampreloxetine (N=110)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Paraparesis (Nervous system disorders) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (2)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (5)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Sciatica (Nervous system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ampreloxetine (N=110)
Urinary tract infection (Infections and infestations) | 8
Headache (Nervous system disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 4

LIMITATIONS AND CAVEATS:
Because the study was terminated early by the Sponsor, the latest scheduled study visit completed by any participant was at Week 98.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/93/NCT04095793/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-13): https://cdn.clinicaltrials.gov/large-docs/93/NCT04095793/SAP_001.pdf